CLINICAL TRIAL: NCT00575341
Title: Dehydroepiandrosterone(DHEA) Substitution in Adolescent and Young Women With Central Adrenal Insufficiency. A Multicenter, Randomised Double Blind Trial
Brief Title: Dehydroepiandrosterone Substitution in Adolescent and Young Women With Central Adrenal Insufficiency
Acronym: DHEA2000
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: PD Dr. med. Gerhard Binder, University-Children's Hospital Tuebingen, Pediatric Endocrinology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DHEA2000 - V18.03.2003; Vorlagen-Nummer BfArM: 4020260
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Adrenal Insufficiency
Keywords: Central Adrenal Insufficiency; DHEA; Pubes
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): substitution of DHEA-hormone, oral, once daily
  Interventions: Drug: Dehydroepiandrosterone
- 2 (Placebo Comparator): substitution of placebo, oral, once daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dehydroepiandrosterone — 25 mg DHEA, oral, once daily
  Arms: 1
Drug: placebo — placebo, oral, once daily
  Arms: 2

SUMMARY:
30 adolescent girls and young women between 13 and 26 years with central adrenal insufficiency and a grand shortage of DHEA are recruit. The clinical trial is double-blind to show that the substitution of the hormone DHEA stimulates secondary hair growth, enhances well being and mood of the patients. It should also normalize the serum content of DHEA, aldosterone and testosterone.

DETAILED DESCRIPTION:
30 adolescent girls and young women between 13 and 26 years with central adrenal insufficiency and a grand shortage of DHEA are recruit. After randomization they either get DHEA or placebo for 12 months daily. The clinical trial is double-blind to show that the substitution of the hormone DHEA stimulates secondary hair growth, enhances well being and mood of the patients. It should also normalize the serum content of DHEA, aldosterone and testosterone.

ELIGIBILITY:
Inclusion Criteria:

* female gender
* age between 13 and 26 Years
* breast developement minimal Tanner stage 3
* serum content of DHEAS less than 400 ng/ml
* central hypocortisolism
* 2 additional pituitary hormon deficiencies (growth hormone, TSH, FSH, LH, prolactin, ADH)
* no scheduled change of the auxilliary medication during the clinical trial

Exclusion Criteria:

* initial diagnosis of a cerebral tumor less than one year
* constitution after cerebral exposure with over 30 gray
* craniopharyngioma with hypothalamic defect syndrome or relapse
* blindness
* mental retardation or psychiatric disorder
* systemic disorder, diabetes mellitus, cardiovascular disease, liver disease requiring treatment
* elevated liver enzyme levels
* pregnancy
* in case of no hypogonadism: no secure contraception

Ages: 13 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2003-10; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Increase of pubes as measured by tanner stage | one year

SECONDARY OUTCOMES:
enhancement in well being and mood by psychometric tests | one year
normalization of the serum content of DHEA, androstanedione and testosterone | one year

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Binder, PD Dr. med., Study Director — Children´s Hospital Tuebingen
Locations (4):
- Germany (4):
  - Universitaere Kinderklinik, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinik für Kinderheilkunde und Jugendmedizin, Tübingen, Baden-Wurttemberg
  - Universitaetskinik für Kinder und Jugendliche, Erlangen, Bavaria
  - Universitaetsklinik und Poliklinik für Kinder und Jungendliche, Leipzig, Saxony

REFERENCES:
- [Background] Miller KK, Sesmilo G, Schiller A, Schoenfeld D, Burton S, Klibanski A. Androgen deficiency in women with hypopituitarism. J Clin Endocrinol Metab. 2001 Feb;86(2):561-7. doi: 10.1210/jcem.86.2.7246. PMID 11158009
- [Background] Young J, Couzinet B, Nahoul K, Brailly S, Chanson P, Baulieu EE, Schaison G. Panhypopituitarism as a model to study the metabolism of dehydroepiandrosterone (DHEA) in humans. J Clin Endocrinol Metab. 1997 Aug;82(8):2578-85. doi: 10.1210/jcem.82.8.4157. PMID 9253337
- [Background] Arlt W, Callies F, van Vlijmen JC, Koehler I, Reincke M, Bidlingmaier M, Huebler D, Oettel M, Ernst M, Schulte HM, Allolio B. Dehydroepiandrosterone replacement in women with adrenal insufficiency. N Engl J Med. 1999 Sep 30;341(14):1013-20. doi: 10.1056/NEJM199909303411401. PMID 10502590
- [Background] Hunt PJ, Gurnell EM, Huppert FA, Richards C, Prevost AT, Wass JA, Herbert J, Chatterjee VK. Improvement in mood and fatigue after dehydroepiandrosterone replacement in Addison's disease in a randomized, double blind trial. J Clin Endocrinol Metab. 2000 Dec;85(12):4650-6. doi: 10.1210/jcem.85.12.7022. PMID 11134123
- [Background] Johannsson G, Burman P, Wiren L, Engstrom BE, Nilsson AG, Ottosson M, Jonsson B, Bengtsson BA, Karlsson FA. Low dose dehydroepiandrosterone affects behavior in hypopituitary androgen-deficient women: a placebo-controlled trial. J Clin Endocrinol Metab. 2002 May;87(5):2046-52. doi: 10.1210/jcem.87.5.8494. PMID 11994339
- [Background] Wit JM, Langenhorst VJ, Jansen M, Oostdijk WA, van Doorn J. Dehydroepiandrosterone sulfate treatment for atrichia pubis. Horm Res. 2001;56(3-4):134-9. doi: 10.1159/000048106. PMID 11847477